CLINICAL TRIAL: NCT00283491
Title: The Effect of a Lactic Acid Fermented Oat Gruel on Iron Absorption in the Proximal and Distal Small Intestine From a Phytate Rich Meal in Healthy Women of Childbearing Age.
Brief Title: The Effect of Lactobacillus Cultures on Iron Bioavailability.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: KF 01-219/03; IHE-KVL-M183
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2005-10

CONDITIONS: Low Iron Stores
Keywords: Iron absorption; Organic acids; Lactobacillus; Probiotic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- A (Active Comparator)
  Interventions: Behavioral: Active Lactobacillus plantarum 299v
- B (Placebo Comparator)
  Interventions: Dietary Supplement: Inactive Lactobacillus plantarum 299v

INTERVENTIONS:
Behavioral: Active Lactobacillus plantarum 299v — 10^11 cfu/meal in 2 meals on 2 consecutive days
  Arms: A
Dietary Supplement: Inactive Lactobacillus plantarum 299v — Inactive form of the active treatment but with the fermentation products in the same concentration
  Arms: B

SUMMARY:
The purpose of this study is to determine the effect of a lactic acid fermented oat gruel on iron absorption in the upper and lower part of the intestine, respectively.

DETAILED DESCRIPTION:
Iron deficiency and low iron stores are prevalent in infants, adolescents, and women of childbearing age in both Western and developing countries. One cause of iron deficiency is the low iron bioavailability from foods, which is partly due to inhibiting factors in the diet, such as phytate and phenolic compounds. A number of single meal studies with lactic acid fermented vegetables and cereals have shown a significant increase in iron absorption in humans. This is believed to be caused mainly by the lactic acid produced during the fermentation process, which conteracts the inhibiting effect of phytate.

A recent study of ours indicate that the increased nonheme iron absorption from a low iron bioavailability meal was due not only to an effect of the lactic acid produced, but also a specific effect of the lactic acid bacteria. As lactic acid bacteria colonizes the entire intestine but mainly the colon it is of interest to determine whether these bacteria can increase iron absorption from the distal part of the intestine since iron absorption normally is believed to be absorbed from the duodenum and most proximal small intestine.

The purpose of this study is therefore to determine the the effect of Lactobacillus plantarum 299v in a lactic acid fermented oat gruel on iron absorption in the proximal and distal small intestine, respectively, in a cross-over design with 18 healthy women of childbearing age, served both fermented oat gruel and pasteurized, fermented oat gruel.

ELIGIBILITY:
Inclusion Criteria:

* serum ferritin in the range 12-30 µg/L
* hemoglobin > 110 g/L

Exclusion Criteria:

* pregnant or lactating
* smoker
* intake of vitamin-, mineral- or other dietary supplements during the study and 2 mo before start
* sports practicing >10h/week
* blood donation during the study and 2 mo before start
* medication
* participation in other isotope studies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-10; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Concentrations of 55-Fe and 59-Fe in blood 18 days after intake in first and second period, respectively (i.e. november and december 2005). | 2 mo

SECONDARY OUTCOMES:
Measurement of serum-ferritin and transferrin receptor in the blood samples before and after each period. | 2 mo

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bukhave, MScD, Study Chair — Department of Human Nutrition, The Royal Veterinary and Agricultural University, Rolighedsvej 30, DK-1958 Frederiksberg C
Locations (1):
- Department of Human Nutrition, The Royal Veterinary and Agricultural University, Frederiksberg C, Denmark